CLINICAL TRIAL: NCT05367362
Title: Efficacy of Minocycline in Improving Neurological Outcomes of Patients Who Undergo Endovascular Revascularization for Acute Ischemic Stroke
Brief Title: Minocycline Efficacy in Improving Neurological Outcome of Patients Who Undergo Endovascular Revascularization for Acute Ischemic Stroke
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study never started, no participants enrolled due to lack of funding
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Adnan H. Siddiqui, Vice Chairman University at Buffalo Neurosurgery, State University of New York at Buffalo
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00006145
Record Dates: First submitted 2022-02-10; First posted 2022-05-10 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Acute Ischemic Stroke
Keywords: Neuroprotection; Acute Ischemic Stroke; Mechanical Thrombectomy; Neuroprotective Drug; Minocycline
MeSH Terms: conditions — Ischemic Stroke; cyclopia sequence | interventions — Minocycline

STUDY DESIGN:
Intervention Model Description: The study will be a prospective, randomized, double- blinded placebo, single center pilot clinical trial.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Patients randomized to minocycline will receive 200mg administered once a day for 21 days. The first dose will be administered in the emergency room or the angiography suite prior to endovascular intervention or within the first two hours of endovascular stroke intervention. If the patient is considered able to swallow as per the routine swallow test, the study drug will be administered orally as intact capsules. If the patient is considered to be at any risk for aspiration or is unable to swallow based on swallowing evaluation, study drug may be started using intravenous route and later switched to oral or via feeding tube as it becomes available.
  Interventions: Drug: Minocyclin
- Control (No Intervention): Patients randomized to control arm will receive look-alike placebo administered once a day for 21 days. The first dose will be administered in the emergency room or the angiography suite prior to endovascular intervention or within the first two hours of endovascular stroke intervention. If the patient is considered able to swallow as per the routine swallow test, the placebo will be administered orally as intact capsules. If the patient is considered to be at any risk for aspiration or is unable to swallow based on swallowing evaluation, placebo may be started using intravenous route and later switched to oral or via feeding tube as it becomes available.

INTERVENTIONS:
Drug: Minocyclin — 200 mg intravenous/oral minocycline hydrochloride for a total of 21 days
  Other Names: Minocycline HCL 200mg Daily (Oral or Intravenous)
  Arms: Intervention

SUMMARY:
The study will be a prospective, randomized, double- blinded placebo, single center pilot clinical trial. Patients with acute ischemic stroke due to large vessel occlusion undergoing endovascular thrombectomy will be included. The treatment group will receive 200 mg intravenous/oral minocycline hydrochloride in addition to endovascular thrombectomy for a total of 21 days. The control group will receive standard medical and endovascular care along with a similar looking placebo. Patients will be randomized to the treatment or control group by the Pharmacy eliminating the selection bias. The patient and evaluator will be blind to the allocation of patients further minimizing the bias. Through randomization we expect to achieve two groups that are comparable in their baseline clinical characteristics.

DETAILED DESCRIPTION:
Overall Design and Rationale for the Study Design The study will be a prospective, randomized, double- blinded placebo, single center pilot clinical trial. Patients with acute ischemic stroke due to large vessel occlusion undergoing endovascular thrombectomy will be included (please see section II - Protocols, for detailed criteria of inclusion and exclusion). The treatment group will receive 200 mg intravenous/oral minocycline hydrochloride in addition to endovascular thrombectomy for a total of 21 days. The control group will receive standard medical and endovascular care along with a similar looking placebo. Patients will be randomized to the treatment or control group by the Pharmacy eliminating the selection bias. The patient and evaluator will be blind to the allocation of patients further minimizing the bias. Through randomization we expect to achieve two groups that are comparable in their baseline clinical characteristics.

Justification of Dose The trial performed by Fagan et al showed minocycline to be safe in patients with acute ischemic stroke at doses as high as 10 mg/kg daily over 72 hours. However, they reported one dose-limiting toxicity being observed at that dose 2. A study by Gordon et al on patients with amyotrophic lateral sclerosis (ALS) showed that minocycline was tolerated well when the dose was at least 300mg daily. However, elevations of nitrogen and liver enzymes were noted over 6-month treatment period 6. On the other hand, when 200-400mg of IV minocycline was used for treatment of infectious disease, 18% of the patients reported at least some adverse effects, half of which were gastrointestinal in nature7.

Considering the above studies, we will administer minocycline at a dose of 200 mg per day for 21 days. This dose is lower than the minimal safe dose reported by Fagan et al2 and does not go over the dose used for ALS or infectious diseases that resulted in some adverse effects. The dose has been used in previous clinical trials on stroke and has proven to be safe and effective. Pharmacokinetic studies have shown that minocycline has a half line approaching 24 hours permitting once daily dosing 2. Unlike previous trials which administered minocycline for 5 days our duration is prolonged i.e., 21 days. This is because of the fact that microglia is one of the main targets for minocycline8, 9. Microglia remain active for several days to weeks after an acute ischemic episode9. Therefore, it may be prudent to continue the drug for that duration.

End of Study Definition A participant will be considered to have completed the study if he or she has completed all phases of the study's last clinical follow up up-to three months. The trial will be concluded after the last participant has completed a 90 day follow up.

II - Protocols Strategies for Recruitment and Retention

Patients will be screened upon presentation to the emergency room with symptoms of acute stroke. All patients considered to have acute ischemic strokes undergo a routine non-contrasted head CT with a subsequent CT perfusion and CT angiogram. A neuroradiologist, a stroke neurologist and a neuroendovascular fellow (with a background training in neurosurgery, neurology or radiology) evaluate these three scans immediately. Based on this immediate screen, patients are triaged to appropriate treatment i.e., intravenous thrombolysis and or intra-arterial in endovascular intervention based on CT angiography and CT perfusion imaging demonstrating salvageable brain tissue.

We will exclude all patients with intracranial hemorrhage. Patients who meet the eligibility criteria for undergoing endovascular revascularization therapy will be presented the option to enroll in the study. An IRB approved informed consent will be obtained from either the patient if he/she can give consent or from an immediate family member or heath care proxy. Patient will then be randomized to intervention or placebo in 1:1 fashion. The randomization will be performed by pharmacy using interactive web response system. The pharmacy will maintain the coding for the patient and intervention given.

Study Population To be eligible for inclusion in the trial patients must meet the following criteria;

1. provision of consent, either by self or authorized representative, willingness and ability to participate in study procedures
2. Acute onset focal neurologic deficit consistent with acute ischemic stroke, or computed tomographic scan consistent with acute cerebral ischemia
3. Age more than 18 years
4. Premorbid Rankin score ≤ 3
5. Treatment with intra-arterial endovascular revascularization methods.
6. Patients should be given first dose of minocycline as soon as possible, latest by 24 hours after the endovascular stroke intervention

All individuals meeting any of the exclusion criteria at baseline will be excluded from study participation:

1. Allergy/ Intolerance to tetracycline antibiotics
2. Pregnant women - positive pregnancy test on admission or known to be pregnant
3. ALT or AST > 3 times the upper limit of normal
4. Serum creatinine > 2 mg/dL
5. Patient is participating in another clinical trial at any time during the duration of the study that could confound the treatment or outcomes of this investigation; and/or
6. Has a severe health condition that may potentially result in death within 6 months.

Study Intervention Administration Minocycline or placebo will be administered to the patients within two hour before or after the endovascular procedure and continued for 21 days. Endovascular revascularization procedure will be performed as planned.

Dosing and Administration

Patients randomized to minocycline will receive 200mg administered once a day for 21 days. The first dose will be administered in the emergency room or the angiography suite prior to endovascular intervention or within the first two hours of endovascular stroke intervention. If the patient is considered able to swallow as per the routine swallow test, the study drug will be administered orally as intact capsules. If the patient is considered to be at any risk for aspiration or is unable to swallow based on swallowing evaluation, study drug may be started using intravenous route and later switched to oral or via feeding tube as it becomes available.

Acquisition and Accountability

Minocycline will be acquired from Kaleida Health Pharmacy. Minocycline and placebo will be prepared and distributed by the pharmacy responsible for providing medicine to the patients in the emergency department and/or angiography suite. Pharmacy shall be responsible for assessing the expiry date of the drug.

Formulation, appearance, packaging, and labeling

Minocycline 200 mg will be mixed with normal saline and given by IV administration, or provided as capsules for the patient to swallow. The placebo will be packaged in a look-alike wrapping. The placebo will have same color and odor. It will not be possible to differentiate it from the placebo which will have same appearance as the drug. The packaging will be performed by the pharmacy.

Product Storage and Stability

The drug will be stored at the room temperature in the pharmacy.

Discontinuation of Study Intervention

If adverse effect is noticed while the patient is admitted, a neurologist will assess the patient and decide on the continuation or discontinuation of the intervention. A form will be filled out by that physician and reported to Dr. Siddiqui who is the PI for this trial. After discharge the patients will be provided a 24 hour emergency line and email of a designated nurse coordinator. The nurse will schedule a visit to the clinic or emergency room. For details on the assessment of adverse events and safety monitoring plan, please see section "Adverse event categorization and safety monitoring".

Participant Discontinuation/Withdrawal from the Study Participants are free to withdraw from participation in the study at any time upon request. An investigator may discontinue or withdraw a participant from the study for the following reason;

1. Pregnancy
2. If the neurologist finds any clinical adverse event, laboratory abnormality, or other medical condition or situation occurs such that continued participation in the study would not be in the best interest of the participant.
3. If the participant meets an exclusion criterion (either newly developed or not previously recognized) that precludes further study participation.
4. Participant unable to receive the intervention for more than 72 hours. The reason for participant discontinuation or withdrawal from the study will be recorded on the Case Report Form (CRF). Subjects who sign the informed consent form and are randomized but do not receive the study intervention may be replaced. Subjects who sign the informed consent form, and are randomized and receive the study intervention, and subsequently withdraw, or are withdrawn or discontinued from the study, will not be replaced.

Lost to Follow Up

A participant will be considered lost to follow-up if he or she fails to return for scheduled three months visit starting from the date of initiation of therapy and is unable to be contacted by the study site staff.

The following actions will be taken if a participant fails to return to the clinic for a required study visit:

* The site will attempt to contact the participant and reschedule the missed visit within a week of missed appointment and counsel the participant on the importance of maintaining the assigned visit schedule and ascertain if the participant wishes to and/or should continue in the study.
* Before a participant is deemed lost to follow-up, the investigator or designee will make every effort to regain contact with the participant (3 telephone calls and a certified letter to the participant's last known mailing address will be dispatched). These contact attempts will be documented in the participant's medical record or study file.
* Should the participant continue to be unreachable, he or she will be considered to have withdrawn from the study with a primary reason of lost to follow-up.

Follow-up and assessment of clinical outcomes A 24h National Institute of Health Stroke Scale (NIHSS) examination will be recorded. MR imaging will be performed as part of routine care. Subsequent follow-up visits will be scheduled at 7-10 days after discharge, 30 days, and 90 days, and include the modified Rankin Scale (mRS) assessing global disability, the Barthel Index assessing instrumental activities of daily living, the NIHSS exam assessing neurologic deficit. The attending neurologist who will be blind to the treatment group will assess the patients on follow up.

Primary outcome The primary study end-point is the degree of disability or dependence at 90 days as assessed by the mRS shift. A global measure of disability, the mRS comprises of seven grades ranging from 0 (no symptoms) to 6 (death). The mRS will be assessed in a formally operationalized manner by use of the Rankin Focused Assessment - Ambulation (RFA-A). The 90-day mRS will be assessed by study personnel certified in the scoring of the mRS using the RFA-A and will be blinded to treatment assignment.

Secondary outcomes

The study secondary end-points are: 1) NIHSS score at 24h; 2) mRS at discharge and 90 days; 3) Barthel Index at 7,30, and 90 days; 4) volume of cerebral infarction as measured by a CT or MRI scan within 72 hours post-procedure. A routine MRI obtained within 72 hours after intervention and at 90 days will be used to calculate the infarct volume. The change in the size of infarct will be also be compared with the infarct size predicted by the pre procedure CT perfusion imaging. Study safety end-points are: 1) all serious adverse events; 2) symptomatic intracranial hemorrhage; 3) any intracranial hemorrhage; 4) myocardial infarction; 5) liver function; 6) mortality and 7) rate of decompressive craniectomies in each group.

NIHSS is a 15-item impairment scale, intended to evaluate neurologic outcome and degree of recovery for patients with stroke. The scale assesses level of consciousness, extraocular movements, visual fields, facial muscle function, extremity strength, sensory function, coordination (ataxia), language (aphasia), speech (dysarthria), and hemi-inattention (neglect)10, 11. The NIHSS was designed to assess differences in interventions in clinical trials, although its use is increasing in patient care as an initial assessment tool and in planning post-acute care disposition10.

The BI was developed in 196512 and later modified by Granger and coworkers13 as a scoring technique that measures the patient's performance in 10 activities of daily life. The BI is considered a reliable disability scale for stroke patients. The items can be divided into a group that is related to self-care (feeding, grooming, bathing, dressing, bowel and bladder care, and toilet use) and a group related to mobility (ambulation, transfers, and stair climbing). The maximal score is 100 if 5-point increments are used, indicating that the patient is fully independent in physical functioning. The lowest score is 0, representing a totally dependent bedridden state.

Adverse events and safety monitoring Adverse event categorization A clinical events committee will validate and categorize the adverse events. This committee will comprise of three expert physicians. Relatedness categories will include: (1) study disease-related: event clearly attributable to underlying disease state with no temporal relationship to the device, treatment, or medication; (2) concomitant disease-related: event attributable to disease other than the study disease with no temporal relationship to the device, treatment, or medication; (3) IV tPA-related: event clearly attributable to IV tPA medication with no temporal relationship to the device or treatment; (4) procedure-related: event has strong temporal relationship to the procedure or treatment of the device implantation or any user handling; (5) Minocycline related: event has a strong temporal relationship to the minocycline and alternate etiology is less likely; (6) other; and (7) unknown.

Patient safety is of paramount importance in this trial, and extensive sets of procedures are in place for monitoring adverse events in the trial. These procedures are as follows:

1. Data Safety Monitoring Board (DSMB). A Data Safety Monitoring Board (DSMB) will meet every 3 months to review the progress of this study (e.g., enrollment, performance) and data on the safety. Before the study begins, the DSMB (in consultation with the study statisticians and principal investigator) will decide on the necessity of an interim analysis, and, if so, the timing of this analysis. Using guidelines established by the committee and the investigators before the study begins, the DSMB may recommend termination of the study if any of the endpoints exceeds pre-established safety thresholds. Additionally, the DSMB may recommend modifications to the protocol if a reversible safety issue is identified. After each meeting, the DSMB Chair will prepare a letter to the study principal investigator, Dr. Adnan Siddiqui, which will describe the safety review that took place at the meeting and that indicates whether any safety concerns exist.
2. Medical Safety Monitor: We have also appointed a safety monitor for the study who will review all adverse events in the study as they occur and consult with the DSMB, if necessary. Before the study begins, the DSMB, after consulting with the study principal investigator and principal statistician will establish a plan for how the monitor will report safety concerns that arise during the trial.
3. Principal Investigator: Dr. Siddiqui will be informed of the DSMB's quarterly assessment of study performance and safety and any other safety issues detected by the Medical Safety Monitor. Additionally, Dr. Siddiqui will monitor any complications, any protocol violations, medication compliance, and risk factor management at the participating sites. If any problems are identified in these areas, Dr. Siddiqui will contact the concerned physicians to rectify the problem.
4. Project Coordinator: Every month, the project coordinator will compile a copy of the adverse event forms to review for events other than primary and secondary endpoints. The purpose of this review is to ensure that these events are recorded and reported and to look for any indications that more serious events may have not been reported.

Drug Related Risks Minocycline is associated with a number of adverse reactions for which patients should be carefully monitored. Our plan to monitor patients according to each adverse reaction described in the drug label is listed below.

Drug Rash with Eosinophilia and Systemic Symptoms (DRESS): during recruitment patients will be screened for any allergic reactions under the use of tetracycline class drugs in the past, either by direct interview with the patient in case of adequate mental status or interview with the family. If allergic reaction occurs during hospitalization, the drug will be discontinued immediately. Patients will also be monitored with complete blood count every 48h to assess for eosinophilia. If patients are discharged home prior to 21 days and continue receiving the drug, instructions will be given to immediately contact medical help in case of rashes, difficulty breathing, pruritus, edema or any other symptoms suggestive of an allergic reaction.

Renal dysfunction: patients will be screened prior to recruitment to exclude those with significant renal function impairment. In those who are enrolled, laboratory assessment of BUN and creatinine levels will be performed every 48h during hospitalization to ensure renal function is under the normal range during treatment period.

Photosensitivity: patients will be oriented to avoid exposure to sun while taking minocycline.

Central nervous system side-effects (lightheadedness, dizziness, vertigo or symptoms): as part of standard of care, patients who undergo endovascular thrombectomy at our institution are constantly monitored by a team including nurses, advanced care practitioners and physicians. Neurological assessment is performed twice a day during rounds to detect any clinical deterioration in these patients.

Hepatotoxicity: patients will be screened prior to recruitment to exclude those with significant liver function impairment and structural compromise. Laboratory assessment of liver enzymes (AST and ALT) and bilirubin will be monitored every 72h during hospitalization.

Laboratory tests mentioned above will also be performed at 7-10 days visit. Protection of Patient Data Research material will include the patient's baseline clinical data (i.e., the patient's history and physical findings, medications), and the results of laboratory tests such as brain CT or MR imaging, CT angiography, electrocardiogram, and blood tests performed to determine the cause of the patient's stroke. Tests done during follow-up as part of routine care such as lipid profile, hemoglobin A1C (if the patient is diabetic), brain CT or MR imaging (if a stroke is suspected), and electrocardiogram (if an MI is suspected) and events that occur as part of the follow-up in the study will be recorded. The results of the 24-48-hours MRI and CTP-CTA acquired as part of the study protocol will be collected. Patient data will be recorded on data forms and it will be stored in a secured database. Information collected during the trial that can be identified with an individual patient will remain confidential and will be disclosed only with the patient's permission. Specific care will be taken so that patient identification will not be disclosed inadvertently in publications that result from this trial (e.g., names on published CT or MRI scans will be covered).

Sample Size Calculation We based our calculation on the clinical trial conducted by Kohler et al4. In order to achieve 80% power at 5% significance level in the Chi-square test, 62 subjects are required for each group to detect a 20% proportion difference of % mRS ≤ 2 between two groups. Anticipating a loss of follow up of 10% we reached a final sample size of 67 per each group.

Statistical analyses A descriptive analysis will performed. Continuous variables with normal distribution will be presented as means and standard deviation while medians and range will be used for skewed data. We will use percentage and proportions to present categorical data. The two groups will be compared for baseline clinical characteristics including age, gender, comorbidities, onset of stroke to intervention delay, NIH score at presentation and pre morbid mRS. We will also compare TICI scores for revascularization in each group. Independent T test will be used to compare continuous variable while chi square will be used to compare categorical data. All the secondary and safety outcomes will also be compared between the groups.

Cochran-Mantel-Haenszel test will be conducted for the shift in Rankin scores. mRS will dichotomized into ≤ 2 and > 2 to estimate the proportion of disability free patients in each group. The odds ratio with 95% confidence interval will be calculated for an mRS ≤ 2 for patients on minocycline. A alpha error of more than 0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

1. provision of consent, either by self or authorized representative, willingness and ability to participate in study procedures
2. Acute onset focal neurologic deficit consistent with acute ischemic stroke, or computed tomographic scan consistent with acute cerebral ischemia
3. Age more than 18 years
4. Premorbid Rankin score ≤ 3
5. Treatment with intra-arterial endovascular revascularization methods.
6. Patients should be given first dose of minocycline as soon as possible, latest by 24 hours after the endovascular stroke intervention

Exclusion Criteria:

1. Allergy/ Intolerance to tetracycline antibiotics
2. Pregnant women - positive pregnancy test on admission or known to be pregnant
3. ALT or AST > 3 times the upper limit of normal
4. Serum creatinine > 2 mg/dL
5. Patient is participating in another clinical trial at any time during the duration of the study that could confound the treatment or outcomes of this investigation; and/or
6. Has a severe health condition that may potentially result in death within 6 months.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
mRS at 90-days | 90 days post op
  The primary study end-point is the degree of disability or dependence at 90 days as assessed by the mRS shift. A global measure of disability, the mRS comprises of seven grades ranging from 0 (no symptoms) to 6 (death). The mRS will be assessed in a formally operationalized manner by use of the Rankin Focused Assessment - Ambulation (RFA-A). The 90-day mRS will be assessed by study personnel certified in the scoring of the mRS using the RFA-A and will be blinded to treatment assignment.

SECONDARY OUTCOMES:
National Institute of Health Stroke Scale (NIHSS) at 24 hours | 90 days post op
  NIHSS at 24 hours will be recorded based on patient's neurologic status by a health care professional to assess stroke severity post-procedure.
  The study secondary end-points are: 1) NIHSS score at 24h; 2) mRS at discharge and 90 days; 3) Barthel Index at 7,30, and 90 days; 4) volume of cerebral infarction as measured by a CT or MRI scan within 72 hours post-procedure. A routine MRI obtained within 72 hours after intervention and at 90 days will be used to calculate the infarct volume. The change in the size of infarct will be also be compared with the infarct size predicted by the pre procedure CT perfusion imaging. Study safety end-points are: 1) all serious adverse events; 2) symptomatic intracranial hemorrhage; 3) any intracranial hemorrhage; 4) myocardial infarction; 5) liver function; 6) mortality and 7) rate of decompressive craniectomies in each group.
mRS at discharge | 24 hours post procedure
  Another secondary outcome measure is the degree of disability or dependence at 90 days as assessed by the mRS scale. A global measure of disability, the mRS comprises of seven grades ranging from 0 (no symptoms) to 6 (death). The mRS will be assessed in a formally operationalized manner by use of the Rankin Focused Assessment - Ambulation (RFA-A).
Barthel Index at 7,30, and 90 days | 7 days, 30 days, and 90 days post procedure
  The Barthel Index (BI) is an ordinal scale used to measure performance in activities of daily living (ADL). Ten variables describing ADL and mobility are scored, a higher number being a reflection of greater ability to function independently following hospital discharge. Time taken and physical assistance required to perform each item are used in determining the assigned value of each item. The Barthel Index measures the degree of assistance required by an individual on 10 items of mobility and self care ADL
Volume of cerebral infarction | 72 hours
  The change in the size of infarct will be compared with the infarct size pre-procedure using CT or MRI within 72 hours post-procedure.
Change in Infarct Volume | 90 days
  A routine MRI obtained at 90 days will be used to calculate the infarct volume. The change in the size of infarct will be also be compared with the infarct size predicted by the pre procedure CT perfusion imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Adnan H Siddiqui, MD PhD, Principal Investigator — University at Buffalo Neurosurgery

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers